CLINICAL TRIAL: NCT03482375
Title: Prospective Evaluation of Residual Bile Duct Stone Detection by Peroral Cholangioscopy That Is Missed With Conventional ERCP and Cholangiogram
Brief Title: Prospective Evaluation of Residual Bile Duct Stone by Peroral Cholangioscopy After Conventional ERCP
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Divyesh Sejpal, Professor of Medicine, Chief of Endoscopy, Northwell Health
Other Study IDs: HS15-0674
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Gall Stones
Keywords: Gall Stones; ERCP; Cholangioscopy
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Stones on POC after ERCP: This is a cohort in which there are no stones seen on Cholangioscopy after ERCP and cholangiogram to treat gall stones.
- Stones seen on POC after ERCP: This is a cohort in which there are no stones seen on Cholangioscopy after ERCP and cholangiogram to treat gall stones.

SUMMARY:
Gallstone disease affects over 20 million Americans. Among patients with gallbladder disease, the prevalence of choledocholithiasis (stones in the bile duct) is estimated to be 10-20%. Endoscopic retrograde cholangiopancreatography (ERCP) is considered the standard of care for removing stones in the bile duct utilizing a variety of conventional methods including biliary sphincterotomy, sphincteroplasty, extraction balloon, retrieval basket, and mechanical lithotripsy. After removal of stones from the bile duct, an occlusion cholangiogram is usually performed to confirm complete bile duct clearance. However, cholangiogram can miss residual stones in 11- 30% of cases - especially in the setting of a dilated bile duct, large stones, severe pneumobilia, juxtapapillary diverticulum, primary sclerosing cholangitis, and after lithotripsy (mechanical, electrohydraulic, or laser). The approach to patients with choledocholithiasis requires careful attention because missed bile duct stones can cause recurrent biliary symptoms, pancreatitis, cholangitis, and has significant cost implication with the need for repeat imaging and/or procedures.

DETAILED DESCRIPTION:
Peroral cholangioscopy (POC) provides direct visualization of the bile duct during ERCP and its benefits are well documented in numerous published studies. POC has been described for therapy of difficult to remove biliary stones utilizing electrohydraulic lithotripsy or laser lithotripsy with success rates of >90%. POC has also been used for evaluation of indeterminate filling defects and to assess for residual stones missed with cholangiogram. In a multicenter study evaluating POC for a variety of indications, 11% (7/66) of patients had bile duct stones identified only by POC that were missed on ERCP. In a study of patients with primary sclerosing cholangitis, 30% (7/23) of patients were found to have stones with POC that were missed with cholangiography. Takao et al. assessed residual bile duct stones found with POC in comparison to balloon-cholangiography; they found that 24% (26/108) of patients had residual stones seen with POC that were missed with balloon-cholangiography.

Although POC has been available for over thirty years, it has not become a widespread technique due to the fact that traditional cholangioscopes are fragile, cumbersome to use, and usually require two endoscopists to perform the procedure. A recent single operator semi-disposable cholangioscope, SpyGlass (Boston Scientific, Natick, Massachusetts), has addressed those concerns and has been shown in a studies to be a useful tool in visualizing the bile ducts and performing therapeutic maneuvers for biliary stones. Both ERCP and Cholangioscopy are standard of care procedures to treat gall stones.

The primary goal of the study is to assess if POC will enhance the diagnostic yield in the detection of residual biliary stones that are missed during conventional ERCP. Residual bile duct stones can especially be seen in the setting of bile duct dilation, history of recurrent abnormal liver function tests, and after lithotripsy (mechanical, electrohydraulic, or laser). Missed biliary stones can lead to recurrent biliary symptoms, pancreatitis, and cholangitis. POC after conventional ERCP can be a useful diagnostic tool to confirm complete extraction of bile duct stones, and thus lead to decreased morbidity and decreased cost by avoiding unnecessary tests and repeat procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receiving ERCP as standard of care for suspected or documented choledocholithiasis as assessed by one or more of the following:

   1. Abnormal imaging on ultrasound, endoscopic ultrasound (EUS), CT scan, or MRCP suggestive of choledocholithiasis
   2. Clinical signs and symptoms suggestive of choledocholithiasis such as jaundice, abdominal pain, pruritis, pancreatitis, and/or cholangitis
   3. Abnormal liver function tests suggestive of choledocholithiasis (eg: serum bilirubin > 1.5 and/or elevated alkaline phosphatase levels)
2. In addition to one or more of the above inclusion criteria, patient must also satisfy one or more of the following:

   1. Mechanical lithotripsy, electrohydraulic lithotripsy, or laser lithotripsy performed for therapy of bile duct stones.
   2. Bile duct > 12mm on prior tests (any portion of duct)
   3. History of recurrent abnormal LFTs with negative cholangiogram.
   4. Positive EUS or MRCP for biliary stones with a negative cholangiogram

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Patients not undergoing ERCP as their standard of care.
3. Patients who had the following surgeries - Billroth II surgery, Roux-en-Y Gastric bypass surgery, and Whipple's surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing ERCP as their standard of care for treatment of their gall stones.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Missed stones found on Cholangioscopy | We will enroll approximately 100 patients over a 2-year period.
  The primary outcome of this study is to assess if digital peroral cholangioscopy (POC) will enhance the diagnostic yield in the detection of residual biliary stones that are missed during conventional ERCP. The primary outcome will be assessed at the time of the procedure (i.e. residual stone seen with POC vs. no residual stone seen with POC). We will enroll approximately 100 patients over a 2-year period. At study completion, the primary outcome measure for all patients will be analyzed and data will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Divyesh Sejpal, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - LIJ Medical Center- NSLIJ Health System, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Everhart JE, Khare M, Hill M, Maurer KR. Prevalence and ethnic differences in gallbladder disease in the United States. Gastroenterology. 1999 Sep;117(3):632-9. doi: 10.1016/s0016-5085(99)70456-7. PMID 10464139
- [Background] Neuhaus H, Feussner H, Ungeheuer A, Hoffmann W, Siewert JR, Classen M. Prospective evaluation of the use of endoscopic retrograde cholangiography prior to laparoscopic cholecystectomy. Endoscopy. 1992 Nov;24(9):745-9. doi: 10.1055/s-2007-1010576. PMID 1468389
- [Background] Lacaine F, Corlette MB, Bismuth H. Preoperative evaluation of the risk of common bile duct stones. Arch Surg. 1980 Sep;115(9):1114-6. doi: 10.1001/archsurg.1980.01380090080019. PMID 7416958
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Awadallah NS, Chen YK, Piraka C, Antillon MR, Shah RJ. Is there a role for cholangioscopy in patients with primary sclerosing cholangitis? Am J Gastroenterol. 2006 Feb;101(2):284-91. doi: 10.1111/j.1572-0241.2006.00383.x. PMID 16454832
- [Background] Itoi T, Sofuni A, Itokawa F, Shinohara Y, Moriyasu F, Tsuchida A. Evaluation of residual bile duct stones by peroral cholangioscopy in comparison with balloon-cholangiography. Dig Endosc. 2010 Jul;22 Suppl 1:S85-9. doi: 10.1111/j.1443-1661.2010.00954.x. PMID 20590779
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] Piraka C, Shah RJ, Awadallah NS, Langer DA, Chen YK. Transpapillary cholangioscopy-directed lithotripsy in patients with difficult bile duct stones. Clin Gastroenterol Hepatol. 2007 Nov;5(11):1333-8. doi: 10.1016/j.cgh.2007.05.021. Epub 2007 Jul 23. PMID 17644045
- [Background] Arya N, Nelles SE, Haber GB, Kim YI, Kortan PK. Electrohydraulic lithotripsy in 111 patients: a safe and effective therapy for difficult bile duct stones. Am J Gastroenterol. 2004 Dec;99(12):2330-4. doi: 10.1111/j.1572-0241.2004.40251.x. PMID 15571578
- [Background] Farrell JJ, Bounds BC, Al-Shalabi S, Jacobson BC, Brugge WR, Schapiro RH, Kelsey PB. Single-operator duodenoscope-assisted cholangioscopy is an effective alternative in the management of choledocholithiasis not removed by conventional methods, including mechanical lithotripsy. Endoscopy. 2005 Jun;37(6):542-7. doi: 10.1055/s-2005-861306. PMID 15933927
- [Background] Chen YK, Pleskow DK. SpyGlass single-operator peroral cholangiopancreatoscopy system for the diagnosis and therapy of bile-duct disorders: a clinical feasibility study (with video). Gastrointest Endosc. 2007 May;65(6):832-41. doi: 10.1016/j.gie.2007.01.025. PMID 17466202
- [Derived] Sejpal DV, Trindade AJ, Lee C, Miller LS, Benias PC, Inamdar S, Singh G, Stewart M, George BJ, Vegesna AK. Digital cholangioscopy can detect residual biliary stones missed by occlusion cholangiogram in ERCP: a prospective tandem study. Endosc Int Open. 2019 Apr;7(4):E608-E614. doi: 10.1055/a-0842-6450. Epub 2019 Apr 12. PMID 30993165

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03482375/Prot_SAP_000.pdf